## Children's Hospital Los Angeles

## CONSENT/PERMISSION/ASSENT¹ TO PARTICIPATE IN A RESEARCH STUDY

# Phase I-II Study of MEK 162 for Children with Low-Grade Gliomas and Other Ras/Raf/ERK Pathway Activated Tumors

#### **Phase II**

| Subject's Name: | |
|-----------------|-------------|
| CHLA#: | Birth Date: |

#### INTRODUCTION

You are invited to participate in a research study conducted by Dr. Nathan Robison, from the Division of Hematology/ Oncology at Children's Hospital Los Angeles (CHLA). This study is being supported by the Neurofibromatosis Clinical Trials Consortium, the Pediatric Low Grade Astrocytoma (PLGA) Foundation, Team Jacks Foundation, Gateway Foundation, The Goldhirsh-Yellin Foundation, Southern California Clinical and Translational Science Institute, Array BioPharma, and the Department of Defense (DOD). You are invited to participate in this study because you have a progressive or recurrent tumor for which no effective standard therapy exists. This study has two parts, a phase I and a phase II. This consent form discusses the phase II part of the study. The phase II part of the study is expected to enroll approximately 90 patients from centers across the country and 5-10 patients from CHLA. Participation in this study is voluntary. Please read the information below and ask questions about anything you do not understand before deciding whether to participate.

#### PURPOSE OF THE STUDY

This study involves treatment of children and adolescents with an experimental drug called MEK162, or binimetinib. This drug has been shown to inhibit (turn off) a molecular pathway called the Ras/Raf/ERK pathway. It does this by blocking the activity of a molecule called MEK1/2. This pathway is abnormally activated (turned on) in some tumors. Inhibiting this pathway may cause some tumors to shrink or to stop growing.

The main purpose of the phase II part of this study is to determine whether MEK162 is able to cause specific tumors in children and adolescents to shrink or stop growing. Other purposes of this study include learning more about the side effects of MEK162 in children, learning how the body handles MEK162 by studying levels of the drug in the blood, and looking for ways to predict how well a tumor will respond to the drug.

<sup>&</sup>lt;sup>1</sup> This form also serves as the permission form for the parent(s) to read and sign. In this case, "You" refers to your child.

#### PROCEDURES

Participation in this research will last up to approximately 2 years. If you volunteer to be in this study, we will ask you to do the following things:

#### BEFORE YOU BEGIN THE STUDY TREATMENT ...

The study doctor will discuss with you your responsibilities as a study participant. You will need to have exams, tests, or procedures to find out if you can receive the study treatment. These exams, tests, or procedures are part of regular care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

#### STUDY DRUG-MEK162

You will take the study drug MEK162 by mouth (swallow a liquid or tablets) 2 times a day for 4 weeks. This 4-week period of time is called a course. The course will be repeated up to 12 times. Each course is numbered in order. You may stay on this study for 12 courses if you do not experience any unacceptable side effects and your tumor does not grow larger. You may continue for an additional 12 courses if your research doctor thinks you are receiving benefit. You can take the study drug with or without food. You will be asked to write down every time you take your study drug in a diary along with any potential side effects. Remember to bring your diary and MEK162 bottles (including empty bottles) with you to all clinic visits. Your research doctor is responsible for reviewing the diary with you at each study visit.

**Research Tests** - The following blood tests are done for research purposes only.

- Pharmacokinetic Blood Samples This involves drawing a small (2 mL each time, or less than half a teaspoon) amount of blood to measure the amount of the study drug in the blood. Most days when these blood samples are drawn, we'll just take one sample. However, on 2 visits during the first course you will have 6 samples drawn over about 6 hours. The total amount of blood drawn over the entire course of the study for pharmacokinetics is approximately 32 mL (a little over 2 tablespoons).
- Biomarker Blood, Urine and Tissue Samples The purpose of the biomarker studies is to help understand whether the drug is acting as expected, and to find out whether results of blood and urine tests can predict how well the drug will work. This involves drawing blood samples (6-16mL, approximately 1-3 teaspoons) and providing your tumor samples to measure the effect of the drug on your tumor. Blood for biomarker studies will be drawn no more than once per month. One blood test will be performed on the first day of the course, 6 hours after a dose of drug. The other blood tests will be performed at the same time as other scheduled blood tests. The maximum total amount of blood drawn over the entire course of the study for the biomarker tests is approximately 68 mL (4 and one half tablespoons). In addition, if able, you will be asked to provide urine in a cup at some study visits.
- Cerebrospinal Fluid Sample (CSF, only collected if clinically indicated)
  If your doctor decides to collect CSF as part of your standard of care, we would like to collet up to 10mL (2 teaspoons) of additional CSF. This CSF sample will only be collected

if you happen to be undergoing the procedure for standard of care purposes. You do not need to undergo this procedure to participate in the study.

## **Target Validation Study (OPTIONAL)**

If you need to have surgery as part of your tumor treatment, you may be eligible to participate in the optional target validation component of the study. If you participate in the target validation component, you will begin taking the study drug 7 to 21 days before your planned surgery. At the time of surgery, part of the tumor that is removed will be set aside and given to researchers for specific tests related to the study. After your surgery, you will start taking the drug again. Your treatment will be the same as for patients on this study who do not participate in the target validation component. You will have the same tests and procedures that are described above.

## **Biorepository (OPTIONAL)**

We would like to store any leftover tissue, blood, urine, and/or CSF samples after analysis at the Dana Farber Cancer Institute for future research use. The future research that will be conducted with the specimens/data will look at what this drug does to the body when given to patients with brain tumors and how the cells in the body express the genes (blue print of DNA). You and your doctor will not be given the results of these research tests because they will have no impact on your care. The results of these research studies may help individuals who receive this drug in the future. Analysis of all tissue and blood samples will be performed at the Dana Farber Cancer Institute. Blood and tissue samples will be identified with a code number and not with your name. You will not be identified directly. You will be assigned a subject ID # which will be used to submit these specimens to Dana Farber Cancer Institute. If you choose to withdraw from the biorepository, please contact your study doctor, and the site staff will notify the Dana Farber Cancer Institute of your withdrawal from the repository. You will be asked if you want to store your leftover samples for future research at the end of the consent form.

#### STUDY CHART

The chart below shows what will happen to you during Course 1 and future treatment courses of treatment. The left-hand column shows the day/week in the course and the right-hand column tells you what to do on that day.

| Course 1 of Treatment | |
|---|---|
| Prior to/On Day 1 | The following procedures are required <u>prior to starting therapy</u> (Course 1, Day 1). These are done as standard of care, but the data collected will be used for research purposes: |
| | <ul> <li>Within 4 weeks of starting treatment:</li> <li>Tumor assessments (MRI scans) to measure the size and shape of your tumor.</li> <li>Eye Exam - you will be seen by an eye doctor. The eye doctor will use drops to cause your pupils (the black part of your eye) to widen so they can see the back of your eyes. The eye doctor will shine a bright light into each eye to see if there are any problems with your eyes.</li> </ul> |

| | <ul> <li>Within 2 weeks of starting treatment: <ul> <li>Medical History</li> <li>Physical Exam, Vital Signs, Height, Weight</li> <li>Blood and urine tests</li> <li>ECG and ECHO (heart tests)</li> </ul> </li> <li>Within 48 hours of starting treatment: <ul> <li>Pregnancy tests (blood or urine) if you are a female of childbearing age. Your pregnancy results will not be shared with your parent(s)</li> </ul> </li> </ul> |
|---|---|
| The following procedures are to be performed on Course 1, Day being done as standard of care, but the data collected will be research purposes: • Medical History • Physical Exam, Vital Signs, Height, Weight • Blood and urine tests | |
| | <ul> <li>Following are being done for research purposes only ("study tests"):</li> <li>Pharmacokinetic Blood Samples (before the first morning dose of MEK162, and at 30-minutes, 1 hour, 2 hours, 4 hours, and 6 hours after that first dose, 2 mL each)</li> <li>Biomarker Blood Sample (16 mL)</li> <li>Tumor Sample (from previous biopsy, if performed)</li> <li>Urine sample</li> <li>Quality of life survey (English and Spanish speakers only)</li> </ul> |
| Day 2 | Pharmacokinetic Blood Sample (2 mL, before the morning dose of MEK162 (for research purposes only) |
| Day 15 | <ul> <li>Blood and urine tests</li> <li>Pharmacokinetic Blood Sample (before the morning dose of MEK162, and at 30-minutes, 1 hour, 2 hours, 4 hours, and 6 hours after that dose) (for research purposes only)</li> </ul> |
| Courses 2-12 | |
| Day 1 of every<br>Course | <ul> <li>Medical History</li> <li>Physical Exam, Vital Signs, Height, Weight</li> <li>Blood and urine tests</li> <li>Pregnancy tests (blood or urine) if you are a female of childbearing age</li> </ul> |
| Day 1 of course 2-4 | Pharmacokinetic Blood Sample (before the morning dose of MEK162 (2 mL, for research purposes only) |
| Day 1 of Course 4 (4-6 hours after dose) | Biomarker Blood Sample (6 mL, for research purposes only) |
| Before Courses 2, 4, and 7 | <ul><li>ECG and ECHO (heart tests)</li><li>Eye Exam</li></ul> |

| | <ul> <li>Tumor assessments (MRI scans) to measure the size and shape of your tumor</li> <li>Biomarker Blood and Urine Sample (10 mL, for research purposes only)</li> <li>Quality of life survey (for research purposes only, English and Spanish speakers only)</li> </ul> |
|---|---|
| Before Course 10 | <ul> <li>Eye Exam</li> <li>ECHO (heart test)</li> <li>Tumor assessment (MRI scan) to measure to size and shape of your tumor</li> </ul> |
| Year 2 (courses 13-24) | |
| Day 1 of Course 13 | • ECG (heart test) |
| Day 1 of Courses 13, 16, 19 and 22 | <ul> <li>Medical History</li> <li>Physical Exam, Vital Signs, Height, Weight</li> <li>Blood and urine tests</li> <li>Pregnancy tests (blood or urine) if you are a female of childbearing age</li> <li>Tumor assessments (MRI scans) to measure the size and shape of your tumor</li> <li>ECHO (heart test)</li> </ul> |
| Day 1 of Courses 13 and 19 | Eye Exam |

#### **End of therapy**

The following procedures are required when you stop taking the study medication. These are done as standard of care, but the data collected will be used for research purposes:

- Medical History
- Physical Exam, Vital Signs, Height, Weight
- Tumor assessments (MRI scans) to measure the size and shape of your tumor.
- ECG and ECHO
- Blood and urine tests
- Pregnancy tests (blood or urine) if you are a female of childbearing age
- Eye Exam

The following procedures will be performed on day 1 of course 13 OR when you top taking the medication, whichever happens sooner:

- Pharmacokinetic and Biomarker Blood Sample (for research purposes only)
- Quality of life survey (for research purposes only, English and Spanish speakers only)

#### • POTENTIAL RISKS AND DISCOMFORTS

The side effects listed below have been seen in adults taking this drug. Children and teenagers taking this drug may have different side effects than the ones shown here. You may experience

other side effects that are not listed below. It is important that you notify your study physician of any new side effects as soon as possible.

#### **Side Effects of MEK162:**

MEK162 is an investigational drug and not all of the side effects are known. Serious side effects, including death, are possible. The long-term effects of MEK162 are also unknown.

Side effects in cancer patients treated with MEK162 (in any treatment group) may include those described below.

## Very Common side effects (greater than 10% incidence)

- Rash, acne or skin irritation including redness, raised bumps, or dryness
- Swelling due to fluid retention or a worsening of pre-existing fluid retention in specific areas of the body. This can occur throughout your body or in specific areas such as your abdomen or arms, legs, hands, feet, face, or eyes.
- An increased value in a lab test called creatine phosphokinase (an enzyme found in the blood that may indicate muscle inflammation or damage or other serious problems if increased)
- Feeling weak, tired, or lacking in energy
- Changes in hair, including hair thinning or change in hair color
- Infection of the skin around the fingernails or toenails
- Muscle weakness. This may affect any part of the body, including neck muscles (resulting in difficulty holding the head up), arms, or legs.
- Anemia (reduction in red blood cells)
- Decreased levels of protein (albumin) in the blood
- Weight gain
- \*Decrease in the heart's ability to pump blood (decreased ejection fraction or left ventricular dysfunction)
- Stomach pain
- Diarrhea
- Nausea
- Vomiting
- Fever
- Increase in lab results that check how well the liver is working
- High blood pressure

#### Common Side effects (1% up to 10% incidence)

- \*Changes in the retina (the light sensing part of the back of the eye), including possible retinal detachment. This may cause blurred or impaired vision.
- Alteration in how things taste or loss of the ability to taste
- Nose bleed
- Blood clots in veins in the legs, in veins of the eyes or in arteries of the lungs
- Changes in heart rhythm
- Dizziness

- Infection of the skin or beneath the skin.
- Skin cracking
- Mouth sores
  - Decreased appetite

## \*Additional information about eye disorders and decreased ejection fraction side effects

Eye disorders: MEK162 has caused mild to moderate visual changes in some adult patients treated with this drug. These changes include swelling and/or inflammation in and around the eyes and changes in the retina. While this type of visual impairment may resolve, there is a risk that the visual changes may continue. Blurred vision and, in some cases, loss of vision may be observed with MEK162. There is the possibility that these changes could affect the activities of your daily life (for example, driving a car or operating machinery). Patients with a history of or current retina blood vessel abnormalities will not be able to participate in this study. All patients will undergo a detailed eye examination at the start of the study. It is important to tell your doctor about any pre-existing eye problems you have and visual changes that occur while taking the study drug as your doctor may decide to change or stop your treatment with the study drug. We do not yet know whether this same side effect may be seen in children and, if so, how frequently.

**Decreased ejection fraction**: A decrease in ejection fraction has been reported in studies with MEK162. This means that the heart's ability to pump blood throughout the body is decreased. This adverse event has also been described with other similar compounds. Your cardiac (heart) function will be evaluated before and during the study. Patients with severe and recent cardiac abnormalities or events should not receive MEK162.

## Rare but important serious side effects seen in patients receiving MEK162 (less than 1%)

- An adult patient taking the study drug experienced acute liver failure (the liver rapidly lost its ability to function normally) leading to death. Due to this event and the observed increase in the value of liver enzymes, your liver function will be evaluated frequently.
- Hypertensive crisis (severe high blood pressure) was described in one study of adult patients treated with MEK162. Increase of blood pressure may be a potential risk when receiving MEK162. Patients at risk for high blood pressure will be monitored closely. If necessary these patients will receive specific treatment for hypertension.
- A severe skin reaction including serious illness with blistering of the skin, mouth, eyes and genitals has been reported in a patient who received MEK162 in combination with another investigational drug (BYL719). It is possible that one of these drugs may have caused this reaction. Please contact your physician immediately in case of such symptoms.
- A small number of patients and subjects in clinical trials developed hives and/or swelling in the throat, also known as angioedema, which can be a sign of an allergic reaction. Your doctor should be notified immediately if you experience tightness in your throat which may be associated with difficulty breathing.
- Severe muscle damage with breakdown of muscle tissue (rhabdomyolysis) which may result in organ damage such as kidney failure.
- Bleeding from the stomach or small intestine, which may be life threatening

## Other possible risks in children

Several children on this study have developed dangerous or life threatening symptoms which have not been seen in adults taking MEK162. It is unclear whether MEK162 caused these symptoms to occur and, if so, how likely they are to happen to other children taking MEK162.

- A small number of children on this study have developed lung infections (pneumonia) and fluid collections around the lung.
- One child on this study developed air within the wall of the intestine. This may be potentially dangerous and needs prompt medical attention.
- One child on this study developed inflammation of the nerves, causing weakness.

#### REPRODUCTIVE RISKS

You should not become pregnant or get a partner pregnant while on this study. There is not enough information to know if the study drug can affect an unborn baby. You should not breastfeed a baby while on this study. You will need to take safety measures to prevent pregnancy (such as not having sexual intercourse or using a hormonal or barrier method of birth control) for the duration of the study. Check with your study doctor about what kind of birth control methods to use and how long to use them. Some methods might not be approved for use in this study.

If you become pregnant or suspect being pregnant during study treatment or within 8 weeks after completing study treatment, you must inform the Study Doctor immediately, and you have to stop ongoing study treatment immediately. You will not be allowed to continue study treatment if you are pregnant. Your Study Doctor will medically follow your pregnancy until delivery to monitor you and your child's safety.

If you get a partner pregnant while in this study, you will be asked to report the pregnancy to the Study Doctor. Consent from your partner will be needed to allow your Study Doctor to medically follow this pregnancy until delivery to monitor the partner's and child's safety.

## DRAWING BLOOD ("VENIPUNCTURE") RISKS

Risks associated with drawing blood are slight, but some risks include: pain, excessive bleeding, fainting or feeling lightheaded, bruising, infection (a slight risk any time the skin is broken), and multiple punctures to locate veins.

#### **SURVEY RISKS**

Certain questions on the quality of life survey may make some people feel uncomfortable. You will be able to stop or skip questions if they make you feel uncomfortable. This survey will only be given to English and Spanish speakers.

#### LOSS OF CONFIDENTIALITY RISKS

There is a possible risk of loss of confidentiality, but standard measures are in place to protect your medical and research information. Please see the "PRIVACY AND CONFIDENTIALITY" section for more information.

#### **UNFORESEEN RISKS**

Since the study medication is investigational, when taken alone or in combination with other medications, there may be other risks that we do not know about and therefore cannot describe. All drugs have potential risk of an allergic reaction, which, if not treated promptly, could become life- threatening. You should tell your study doctor about any side effect or new health problems that develop while you are participating in this study.

#### ANTICIPATED BENEFITS TO SUBJECTS

The main purpose of phase II clinical trials (like this study) is to test the safety and effectiveness of the treatment. In these types of studies, researchers collect information on side effects that happen in patients and the way your tumor responds to the treatment.

It is possible that the treatment may cause your tumor to shrink or to stop growing; however, the likelihood that this will happen in your tumor is unknown.

#### ANTICIPATED BENEFITS TO SOCIETY

This study may help us learn more about the study drug, MEK162, and about how it works. This study may help us to learn about your tumor. It may help us to improve treatment for children and adolescents with tumors like yours in the future.

#### ALTERNATIVES TO PARTICIPATION

The alternatives to participating in this research study include:

- Other standard treatments. These will vary depending on your specific disease and what treatment(s) you have already received.
- Treatment on a different clinical research study.
- No treatment for your tumor.

Please ask questions about all of your treatment options before deciding whether to participate in this research.

### FINANCIAL OBLIGATION

You and your insurance company will not be charged for the study drug (MEK162) and tests done for research purposes only.

This study includes procedures that are also a part of the standard treatment of your disease. The cost of these procedures will be billed to your insurance or other third-party payer. The cost of treating any side effects of this treatment will also be billed to your insurance or other third-party payer . You may be responsible for any co-pays or deductibles.

Your family is responsible for other costs that may result from your participation in the study, such as time off work, carfare, baby sitter fees, food purchased while at the hospital, etc.

## • EMERGENCY CARE AND COMPENSATION FOR INJURY

The Investigators and CHLA, Department of Defense, Array BioPharma Inc., and the Neurofibromatosis Consortium have made no provision for monetary compensation in the event of injury from the research, and in the event of such injury, treatment will be provided but is not free of charge.

It is important that you promptly tell the study doctor if you feel that you have been injured because of taking part in this study. You can tell the study doctor in person, or call them at 323-361-2121. If you are injured or become ill as a direct result of participating in this study, CHLA will provide necessary medical treatment. The costs of treatment will be billed to you or your insurer like other medical costs. CHLA has no program to provide you with any additional compensation as a result of any injuries. You do not waive any liability rights for personal injury by signing this form.

#### PRIVACY AND CONFIDENTIALITY

Members of the research team and, if appropriate, your physicians and nurses will know that you are a research subject. All results will be kept confidential but may be made available to you and/or your physician, if you wish. No information about you or provided by you during the research will be disclosed to others without your written permission, except:

- if necessary to protect your rights or welfare (for example, if you are injured and need emergency care); or
- if required by law (i.e., child or elder abuse, harm to self or others, reports of certain infectious diseases).

When the results of the research are published or discussed in conferences, no information will be included that would reveal your identity.

Authorized representatives of the Food and Drug Administration (FDA), the Department of Health and Human Services (if applicable), governmental agencies in other countries where the study drug may be considered for approval, the Pediatric Low Grade Astrocytoma Foundation, Team Jacks Foundation, the supplier of the drug being tested (Array BioPharma) and its authorized agents, the CHLA Institutional Review Board (IRB), the Department of Defense (DOD), and the medical monitor may need to review records of individual subjects. A Data and Safety Monitoring Board (DSMB), a research monitor and a site monitor will be reviewing the data from this research throughout the study. As a result, they may see your name.

The doctors at Children's Hospital Los Angeles will review the MRIs of patients on this study. Your MRI will be coded with a unique identifier (a specific study ID number given only to you) by the research staff. Only the coded MRI will be shared with Children's Hospital Los Angeles. They will not see your name or have access to your medical records.

Because this study involves the treatment of a medical condition, a copy of this form will be placed in your medical record. This will allow the doctors that are caring for you to obtain information about what medications or procedures you are receiving in the study and treat you appropriately.

#### • PARTICIPATION AND WITHDRAWAL

Your participation in this research is VOLUNTARY. Your choice about whether or not to participate will have no effect on your care, services, or benefits at Children's Hospital Los Angeles. If you agree to participate, but later decide to withdraw from this study, you may do so without affecting your rights to health care, services, or other benefits at Children's Hospital Los Angeles. Please contact the Principal Investigator if you wish to withdraw from the study.

## • CONSEQUENCES OF WITHDRAWAL

It is important to tell the research doctor if you are thinking about stopping so your research doctor can evaluate the risks from stopping the drug, MEK162. In some cases, the abrupt stopping of a drug can have risks in itself. Another reason to tell your research doctor that you are thinking about stopping is to discuss what follow-up care and testing could be most helpful for you.

#### WITHDRAWAL OF PARTICIPATION BY THE INVESTIGATOR/SPONSOR

The investigator may withdraw you from participating in this research if necessary to protect your health or if other situations arise that make it necessary to do so. Your participation in this study may be terminated by the investigator and/or sponsor, without your consent, for any of the following reasons:

- If you fail to follow the investigator's instructions including not completing the procedures required by the study and/or are unable or unwilling to come for the required doctor visits including any required follow-up visits
- If you experience a serious and unexpected side-effects that may require evaluation.
- If you experience side effects that are considered to outweigh benefits of your participation.
- If your disease gets worse while on this treatment.
- If the investigator feels it is in the best interest of your health and welfare.
- If you become pregnant while on study
- If you begin another treatment or begin taking any other medications that are not allowed during the study.

The investigator, Dr. Nathan Robison, will make the decision and let you know if it is not possible for you to continue. The decision may be made either to protect your health and safety, or because it is part of the research plan that people who develop certain conditions may not continue to participate.

#### NEW INFORMATION

If there is significant new information found during the course of the study or the research plan is changed in a way that might affect your decision to continue participating in the study, you will be informed and your consent to continue participating in the study may be requested.

#### HOW TO OBTAIN INFORMATION

Daytime, Monday through Friday, 8:00 A.M. through 4:30 P.M. you may call Dr. Robison at 323-361-2121.

Evenings, nights, weekends, or holidays you may call the hospital number, 323/660-2450 and ask for the Oncology Service doctor on-call.

If you have non-urgent questions about the research, please call Dr. Nathan Robison, Monday through Friday, 8:00 A.M. through 4:30 P.M.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### FINANCIAL INTEREST OF THE INVESTIGATOR

Funding for this research study is provided by the Pediatric Low Grade Astrocytoma (PLGA) Foundation, Gateway Foundation, Southern California Clinical and Translational Science Institute, The Goldhirsh-Yellin Foundation, Team Jacks Foundation, and the Department of Defense (DOD). The amount of funding is based upon the number of research subjects enrolled. If your physician is an investigator for this study, he/she is interested in both your healthcare and the conduct of this research. You are not under any obligation to participate in a research study conducted by your physician.

#### RIGHTS OF RESEARCH SUBJECTS

You may withdraw from this study at any time and discontinue participation without penalty. You are not waiving any legal claims, rights, or remedies because of your participation in this research study. If you have questions regarding the rights of research subjects or if you have complaints or concerns about the research and cannot reach the Principal Investigator; or just want to talk to someone other than the Investigator, you may call Children's Hospital Los Angeles, Human Subjects Protection Program office at (323) 361-2265.

#### **OPTIONAL RESEARCH STUDIES**

You may take part in these additional studies if you want. You can still be a part of the main study even if you say "no" to taking part in any of these additional studies. You can say "yes" or "no" to each of the following studies. Please provide your initials beside your decision for each study.

#### TARGET VALIDATION STUDY

You may be eligible to participate in the Target Validation component of the study if your doctor has recommended that you undergo surgery to remove part of your tumor. By marking "Yes" below, you agree to participate in the Target Validation component of the study, which will involve beginning the study drug 7 to 21 days before your planned surgery. You also agree to have a portion of the tumor given to researchers for specific tests related to this study. This component of the study is optional. You may initial "No" or "N/A" and still participate in the rest of the study.

| Yes | No | [for subject to complete, if the subject is 14 years or older] |
|---|---|---|
| Yes | No | [for parent to complete, if subject is a minor] |
| N/A [Not | applicable: n | o surgery planned] |
| | ce regarding | if left-over BLOOD samples can be <b>stored for future</b> nents and conditions, and ways to prevent these conditions: |
| Yes | No | [for subject to complete, if the subject is 14 years or older] |
| Yes | No | [for parent to complete, if subject is a minor] |
| • | | if left-over TUMOR TISSUE samples can be <b>stored for</b> s, treatments and conditions, and ways to prevent these |
| Yes | No | [for subject to complete, if the subject is 14 years or older] |
| Yes | No | [for parent to complete, if subject is a minor] |

# SIGNATURE OF RESEARCH SUBJECT (If the subject is 14 years or older)

Your signature below indicates

- You have read this document and understand its meaning;
- You have had a chance to ask questions and have had these questions answered to your satisfaction;
- You consent/assent to your participation in this research study; and
- You will be given a signed copy of this form.

| Print Name of Subject | |
|---|---|
| Signature of Subject | Date |
| SIGNATURE OF PARENT(S)/LEGA | L GUARDIAN(S) (If the subject is a minor) |
| Your signature(s) below indicates | |
| <ul> <li>You have read this document and under</li> </ul> | erstand its meaning; |
| <ul> <li>You have had a chance to ask question<br/>satisfaction;</li> </ul> | as and have had these questions answered to your |
| <ul> <li>You agree to your child's participation</li> </ul> | in this research study; |
| <ul> <li>You will be given a signed copy of this</li> </ul> | s form. |
| Print Name(s) of Parent(s)/Legal Guardian(s) | |
| Signature of Parent/Legal Guardian | Date |
| Signature of Parent/Legal Guardian | Date |
| SIGNATURE OF INDIVI | DUAL OBTAINING CONSENT |
| | d/or the subject's parent(s)/legal guardian(s) and |
| nave answered all of their questions. I believe described in this document and freely give con | that they understand all of the information |
| Print Name of Individual Obtaining Consent | |
| Signature of Individual Obtaining Consent | Date |

## **SIGNATURE OF WITNESS (if applicable)**

Your signature below indicates:

- I was present for the entire consent conference;
- The information in the consent document and any other written information was accurately explained to the subject and/or the subject's parent(s)/legal guardian(s);
- The subject and/or the subject's parent(s)/legal guardian(s) had an opportunity to ask questions and those questions were answered; and
- The subject and/or the subject's parent(s)/legal guardian(s) voluntarily signed the consent/permission/assent form in my presence.

| Print Name of Witness | |
|---|---|
| Signature of Witness | Date |
| Study Team Instructions: Only complete the severbal assent was obtained from the subject or | ection below if assent is required, and either only assent was not obtained from the subject. |
| Please check appropriate box and sign below | |
| The undersigned, from the subject. | , hereby certifies that verbal assent was obtained |
| Assent was not obtained from the subject. (Please state the reason. Examples include: subject is an infant; subject is comatose; subject lacks cognitive abilities to understand the information; etc.) | |
| Date: | |
| Time: Signature | |

Routing of signed copies of the form:

- 1) Give to the subject if at least 14 years old (copy)
- 2) Give to the parent/legal guardian if subject is a minor (copy)
- 3) Place in the CHLA Medical Record (copy)
- 4) Place in the Principal Investigator's research file (original)